CLINICAL TRIAL: NCT04588285
Title: A Clinical Trial to Demonstrate Clinical Efficacy on Cognitive, Neuropsychiatric and Functional Outcomes of Ambroxol in New and Early Patients With Prodromal and Mild Dementia With Lewybodies
Brief Title: Ambroxol in New and Early DLB, A Phase IIa Multicentre Randomized Controlled Double Blind Clinical Trial
Acronym: ANeED
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Fonna (Other)
Collaborators: Klinbeforsk (Other); Helse-Bergen HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3.3 Date: October 1st 2023
Record Dates: First submitted 2020-08-26; First posted 2020-10-19 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Dementia With Lewy Bodies
Keywords: Cognitive; Neuropsychiatric; Functional Outcomes; New and Early Patients; Prodromal; Mild Dementia; Lewybodies
MeSH Terms: conditions — Lewy Body Disease | interventions — Ambroxol

STUDY DESIGN:
Intervention Model Description: Each participant will receive 5 intra-participant dose escalations at 60 mg TID (day 1-7), 120 mg TID (day 8-14), 315 BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550) with ambroxol or placebo for the duration of 18 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded phase (placebo or ambroxol) will last for 18 months and an open extension with ambroxol will be offered to all participants for one additional year. Randomisation to placebo or ambroxol will be done by the system Viedoc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ambroxol (Experimental): Oral ambroxol medication, from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 mg BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)).
  Interventions: Drug: Ambroxol
- Placebo (Experimental): Oral placebo medication, from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 mg BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambroxol — Oral ambroxol medication (60 mg) from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 mg BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)
  Other Names: Mucosolvan
  Arms: Ambroxol
Drug: Placebo — Oral placebo medication (60 mg) from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 mg BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)
  Arms: Placebo

SUMMARY:
This is a confirmatory investigational medicinal product (IMP) study to investigate the effects on cognition, functional decline and on neuropsychiatric symptoms of the Glucocerebrosidase (GCase) enhancing chaperone ambroxol in participants diagnosed with prodromal and early dementia with Lewybodies (DLB).

DETAILED DESCRIPTION:
Participants will be recruited through established network of Norwegian Memory Clinics. Patients will be randomised to ambroxol with proven effect on the lysosomal and glucocerebrosidase pathology in DLB or placebo. The randomization will be stratified based on APOE e4 and on the concentration of A-beta in CSF. The frequency of GBA genotypes in the active treatment and placebo groups will be calculated at study end. The blinded phase will last for 18 months and an open extension with ambroxol will be offered to all participants for one additional year. The primary outcomes will be cognition, global function, disease stage, progression, and neuropsychiatric symptoms. Secondary outcomes will be on sleep disturbances, falls, fluctuations and parkinsonism, and exploratory outcomes will be impact on the potential biomarkers for drug effects defined as qEEG, DaTSCAN, MRI and α-synuclein in CSF. One hundred and eighty participants will be recruited in total. Each participant will orally self-administer or administer by a caregiver ambroxol or placebo at 5 intra-participant dose escalations at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)).Participants will be subjected to clinical and laboratory assessments to assess the safety, tolerability effects of ambroxol on blood biomarkers and MRI, DaTSCAN, ECG, EEG and lumbar puncture. Each participant will undergo 8 hospital visits and 16 telephone visits for the blinded phase of the study during the first 18 months. Hospital visits will additionally include 1 or 2 screening appointments within 60 days of Day 1 hospital visit (at which participants will receive the first dose of ambroxol), followed by visits at week 4, week 8, week 24, week 36, week 52, month 15 and month 18. Participants will receive a telephone call 3 days after lumbar puncture to record any complaints. Participants will receive 16 telephone calls to record any drug related adverse events in between hospital visits, between 1-3 days before and after each dose escalation (day 1, 8, 15, 22 and 29, week 12,16, 20, 28, 32, 40, 44, 48 and month 13, 14, 16 and 17). All participants will be offered treatment with the IMP for 12 additional months from month 18 - month 30.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female.
2. Age ≥ 50 and ≤ 85 years of age.
3. Confirmed diagnosis of Dementia with Lewy Bodies (DLB) or Mild Cognitive Impairment in DLB (DLB-MCI).
4. MMSE score>=15
5. Able and willing to provide informed consent prior to any study related assessments and procedures at screening visit 1.
6. Capable of complying with all study procedures.
7. Willing to provide blood samples for genetic analyses of APOE and GBA.
8. Willing and able to self-administer or administer by a caregiver oral ambroxol medication, from day 1 to study end (at 60 mg TID (day 1-7), 120 mg TID (day 8- 14), 315 BID (day 15-21), 315 mg TID (day 22-28) and 420 mg TID (day 29-550)).
9. Able to travel to the participating study site.
10. A female participant is eligible to participate if she is of:

    Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 consecutive months of spontaneous amenorrhea, at least 6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) or post tubal ligation. In questionable cases, menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 25.8 - 134.8 IU/L and oestradiol < 201 pmol/l at entry.

    Women of child-bearing potential must use accepted contraceptive methods (listed below), and must have a negative serum at screening visit 1 and urine pregnancy tests at subsequent visits if applicable. An additional pregnancy test will be performed, and results obtained, prior to administration of the first dose of ambroxol.
11. A female participant is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 consecutive months of spontaneous amenorrhea, at least 6 weeks post-surgical bilateral oophorectomy (with or without hysterectomy) or post tubal ligation. In questionable cases, menopausal status will be confirmed by demonstrating levels of follicle stimulating hormone (FSH) 25.8 - 134.8 IU/L and oestradiol < 201 pmol/l at entry.

Women of child-bearing potential must use accepted contraceptive methods (listed below), and must have a negative serum at screening visit 1 and urine pregnancy tests at subsequent visits if applicable. An additional pregnancy test will be performed, and results obtained, prior to administration of the first dose of ambroxol.

Exclusion Criteria:

1. Current treatment with anticoagulants (e.g. warfarin) that might preclude safe completion in the opinion of the Investigator.
2. Current use of investigational medicinal product or participation in another interventional clinical trial or who have done so within 30 days prior to the first dose in the current study.
3. Exposure to more than three investigational medicinal products within 12 months prior to the first dose in the current study;
4. Confirmed dysphagia that would preclude self-administration of ambroxol up to 6 tablets daily for the duration of day 1 to day 550/Month 18.
5. Significant known lower spinal malformations or other spinal abnormalities that would preclude lumbar puncture.
6. History of known sensitivity to the study medication, ambroxol or its excipients (lactose monohydrate, granulated microcrystalline cellulose, copovidone and magnesium stearate) in the opinion of the investigator that contraindicates their participation.
7. History of known rare hereditary disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
8. History of illegal substance abuse, drug abuse or alcoholism in the opinion of the Investigator that would preclude participation in the study.
9. Donation of blood (one unit or 350 ml) within three months prior to receiving the first dose of the study drug.
10. Pregnant or breastfeeding; All participants of child bearing potential in the opinion of the Investigator that would preclude participation in the study and who do not agree to use double-barrier birth control or abstinence while participating in the study and for two weeks following the last dose of study drug;
11. Any clinically significant or unstable psychiatric, medical or surgical condition that in the opinion of the PI or PI-delegated clinician may put the participant at risk when participating in the study or may influence the results of the study or affect the participant's ability to take part in the study, as determined by medical history, physical examinations, electrocardiogram (ECG), or laboratory tests.

    Such conditions may include:
    1. Impaired renal function
    2. Moderate/Severe hepatic impairment
    3. A major cardiovascular event (e.g. myocardial infarction, acute coronary syndrome, decompensated congestive heart failure, pulmonary embolism, coronary revascularisation that occurred within 6 months prior to the screening visit.
    4. Major depression, delirium or psychosis not related to DLB.
    5. Metastatic cancer or terminal illness.
12. Planned major surgery or other major treatments during study period that will interfere with study-obligations.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence, nature and severity of AE's and SAE's from baseline. | All patient visits including phonecalls trough study completion, planned duration 18 months
  Change in the number of participants with AE's and SAE's.
Change in the number of participants with treatment discontinuations and study discontinuation due to AEs from baseline. | All patient visits including phonecalls trough study completion, planned duration 18 months
  Change from baseline in the number of participants with treatment and/or study discontinuation will be used to demonstrate safety and tolerability
Change in the number of participants with electrocardiogram (ECG) abnormalities. | Through study completion at the following visits: Screening, Baseline, week 4, week 24, week 36, week 52, month 15, and month 18.
  Including QTc interval.
Change in blood analyses from baseline over time abnormalities. | Through study completion at the following visits: Screening, week 4, week 8, week 24, week 36, week 52, month 15, and month 18.
  Change from baseline in number of participants with abnormal changes in clinical laboratory blood tests from baseline over time for safety.
Change in MMSE-NR3 (Mini Mental Status Examination, Norwegian revised version) over time. | Through study completion at the following visits: Screening, week 24, week 36, week 52, Month 18.
  To confirm the effect of the IMP ambroxol in participants diagnosed with DLB measured by a defined battery of cognitive tests defining MMSE-NR3 as the primary outcome.
  The MMSE-NR3 is a screening test for cognitive impairment that spans the visuospatial/executive, naming, memory, attention, language, delayed recall and orientation domains (score range from 0 to 30 points).
ADCS-CGIC (Clinician's Global Impression of Change) | Through study completion at the following visits: Screening, week 24, week 36, week 52, month 18.
  To confirm the effect of the IMP Ambroxol on the rate of functional decline in DLB.
Change in CDR-SB (Clinical Dementia Rating-Sum of Boxes). | Through study completion at the following visits: Screening, week 24, week 36 week 52, Month 18.
  Measure Rate of decline from screening to study completion at month 18 using CDR-SB.
Change NPI (neuropsychiatric inventory) | Through study completion at the following visits: Screening, week 24, week 36, week 52, month 18.
  To confirm the effect of the IMP Ambroxol on neuropsychiatric symptoms in DLB from screening to study completion at month 18 by using NPI.
  The NPI is a semistructured clinician interview of caretakers in which the severity and frequency of disturbance in 12 symptom domains is rated. The scoring reflects not only the effect on the patient, but also the extent to which the symptom causes distress in the caregiver.
  Score 0-144. The higher the score the more disease progression.
GDS (geriatric depression scale) - 15 items | Through study completion at the following visits: Screening, week 24, week 36, week 52, month 18.
  To confirm the effect of the IMP Ambroxol on neuropsychiatric symptoms in DLB from screening to study completion at month 18 by using GDS.
  The Geriatric Depression Scale (GDS) is a 15-item self-report assessment used to identify depression in the elderly. A high score usually always indicates depression and more severe depression.

SECONDARY OUTCOMES:
Mayo Sleep Questionnaire (MSQ). | Through study completion at the following visits: Screening, week 24, week 36, week 52, Month 18.
  To confirm the effect of The IMP Ambroxol in DLB measured on MSQ for evaluating sleep disturbances.
  MSQ is developed and validated in English version to detect Rapid Eye Movement - (REM) Sleep Behavior Disorder - (RBD) and several other sleep disorders in people with dementia and Parkinson's disease. RBD is part of the diagnosis of dementia with Lewy bodies.
  No score - only yes/no questions.
Mayo Fluctuation Scale (MFS) | Through study completion at the following visits: Screening, week 24, week 36, week 52, Month 18.
  To confirm the effect of The IMP Ambroxol in DLB measured on MFS for evaluating fluctuations.
  The Mayo Fluctuations Scale is a short questionnaire that evaluates cognitive fluctuation.
  Three or four points shows cognitive fluctuation. Scale 0-4.The higher the score the more disease progression
Unified Parkinson Disease Rating Scale (UPDRS-III) | Through study completion at the following visits: Screening, week 8, week 24, week 36, week 52, Month 18.
  To confirm the effect of The IMP Ambroxol in DLB measured on UPDRS-III for evaluating Parkinsonism.
  The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease. Following the UPDRS scores over time provides insight into the patient's disease progression.
  Scale 0-138 points. The higher the score the more disease progression
Number of falls and related injury | Through study completion at the following visits: Screening, week 24, week 36, week 52, Month 18.
  To confirm the effect of The IMP Ambroxol in DLB measured on questions evaluating number of falls and related injury.

CONTACTS AND LOCATIONS:
Overall Officials: Arvid Rongve, Phd, Principal Investigator — arvid.rongve@helse-fonna.no
Locations (1):
- Helse Fonna, Haugesund, Norway

IPD SHARING:
Plan to Share IPD: No
All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.

REFERENCES:
- See also: Rongve, A., et al. Demens med Lewylegemer- utredning og behandling. 2017 — https://www.helsebiblioteket.no/fagprosedyrer/ferdige/demens-med-lewylegmer-utredning-og-behandling
- See also: Aarsland, D. MULTI-CENTRE COHORT-STUDIES IN LEWY-BODY DEMENTIA. 2015 — http://www.neurodegenerationresearch.eu/wp-content/uploads/2015/10/JPND-Report-Aarsland.pdf